CLINICAL TRIAL: NCT05432154
Title: Efficacy and Safety of a Novel Silicone Wound Dressing for the Management of Atrophic Vaginitis
Brief Title: An Innovative Silicone Wound Dressing for the Management of Atrophic Vaginitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stratpharma AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPAMG01
Record Dates: First submitted 2022-06-20; First posted 2022-06-27 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Atrophic Vaginitis
MeSH Terms: conditions — Atrophic Vaginitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment arm (Experimental): Patients apply 7-0940 at least 2 times daily for 3 months.
  Interventions: Device: Film forming silicone gel (7-0940)

INTERVENTIONS:
Device: Film forming silicone gel (7-0940) — Film forming silicone gel (7-0940) is an innovative gel that forms a full contact, flexible wound dressing for supporting mucosal conditions of the genital, rectal and perineal areas.
  Film forming silicone gel (7-0940) is a semi-occlusive, non-resorbable, self-drying and transparent gel.
  Film forming silicone gel (7-0940) may be directly applied to dry, wet, cracked and sensitive mucosal tissue.
  Film forming silicone gel (7-0940) gel is bacteriostatic and inert. It contains no alcohols, parabens or fragrances.

SUMMARY:
The objective of the study is to determine the efficacy of 7-0940 in the management of atrophic vaginitis in female patients

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent
* Diagnosed acute or chronic Atrophic Vaginitis
* Controlled disease, or uncontrolled disease that did not respond to standard therapy with HRT

Exclusion Criteria:

* Unable to provide informed consent
* Patient unable to apply topical device
* Allergy or intolerance to ingredients or excipients of the formulation of studied products
* Currently on HRT (orally or topically)
* Currently on corticosteroid treatment

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Patient-reported Vulvar Quality of Life | 3 months
  Vulvar Quality of Life Index

SECONDARY OUTCOMES:
Patient-reported symptoms | 3 months
  Likert scales to measure:
  * Pruritus/itchiness
  * Tender/sore
  * Swelling
  * Dryness
  * Burning of skin
  * Dyspareunia
  * Stinging with urination/clothes
  * Defecating pain/burning
Severity of overall condition | 3 months
  Clinician-rated severity of atrophic vaginitis
Product rating | 3 months
  Likert scale for product rating by the patient

CONTACTS AND LOCATIONS:
Locations (1):
- Orange Coast Women's Medical Group, Laguna Hills, California, United States

IPD SHARING:
Plan to Share IPD: No